CLINICAL TRIAL: NCT04388306
Title: Functional Performance of Shoulder After Arthroscopic Rotator Cuff Repair and Investigation of Performance Related Factors
Brief Title: Shoulder Functional Performance After Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Beyza Yazgan Dagli, Research Assistant, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-BYD-01
Record Dates: First submitted 2020-05-06; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Thirty-two participants with undergone arthroscopic Rotator Cuff repair
  Interventions: Other: Shoulder Performance Test- Functional Impairment Test-Head and Neck, Shoulder, Arm (FIT-HaNSA)
- Control Group: Thirty-two healthy participants
  Interventions: Other: Shoulder Performance Test- Functional Impairment Test-Head and Neck, Shoulder, Arm (FIT-HaNSA)

INTERVENTIONS:
Other: Shoulder Performance Test- Functional Impairment Test-Head and Neck, Shoulder, Arm (FIT-HaNSA) — Participants were evaluated with all tests, respectively. To eliminate the fatigue factor, 5 minutes breaks were given after each test.
  Other Names: Shoulder Functionality-Modified Constant Murley Score; Scapular Endurance-Scapular Muscle Endurance Test; Strength-Total Upper Extremity Muscle Strength

SUMMARY:
Rotator Cuff (RC) injuries are a progressive clinical condition that starts with an acute tendonitis, continues with partial thickness rupture and results in a full thickness rupture in the advanced period.

Arthroscopic RC repair is effective in the acute RC ruptures treatment caused by traumatic events. In the acute period after arthroscopic RC repair, shoulder joint range of motion (ROM), muscle strength and shoulder functionality are decreased and daily activities are adversely affected. In the long-term, many studies have reported that these symptoms gradually decreaced.

Many studies investigating postoperative treatment of RC rupture have mostly focused on parameters such as postoperative pain, functionality, muscle strength, ROM and quality of life.Evaluation of these clinical parameters is necessary for patient follow-up in the early period. However, it is unclear whether the biomechanical etiologic factors continue that lead to RC rupture in the advanced period after surgery.

Therefore, the objective of this study was functional performance of shoulder after arthroscopic Rotator Cuff repair and ınvestigation of performance related factors.

DETAILED DESCRIPTION:
Design: observational Cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* With the same RC surgical procedure and technique,
* With acromioplasty and/or tenodesis with RC repair,
* Undergoing arthroscopic RC repair from the upper extremity of the dominant side,
* Having completed the 12th week after surgery,
* Performing 90° and above active shoulder elevation movement

Exclusion Criteria:

* Having undergone revision surgery or previous shoulder surgery, a history of fracture of the upper extremity
* Having undergone surgery causing limitation of motion in the spine,
* Having a neurological and/or vestibular and/or rheumatologic disease,
* Participants with diabetes mellitus, hypertension, cardiovascular and chronic respiratory disease that may cause problems during the test

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group consists of participants with undergone arthroscopic RC repair at Bolu Abant İzzet Baysal University, Department of Orthopedics and Traumatology.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Functional Impairment Test-Head and Neck, Shoulder, Arm (FIT-HaNSA) | Three months
  FIT-HaNSA is a test battery consisting of 3 tasks simulating overhead work and lifting activities designed to evaluate the shoulder functional performance.

SECONDARY OUTCOMES:
Modified Constant Murley Score | Three months
  Shoulder functionality was analyzed by using the MCMS evaluating pain, daily living activities, ROM and strength. Pain was evaluated by visual analog scale and ROM by goniometer. The force in the shoulder abduction position was measured with the Digital analyzer defined by the spring balance technique.
Scapular Muscle Endurance Test | Three months
  The scapular muscle endurance test evaluate the endurance of the serratus anterior and the trapezium muscles.
Total Upper Extremity Muscle Strength | Three months
  Total upper extremity muscle strength was evaluated with Jamar hand dynamometer. Grip strength is considered to be a valid value of TUEMS. The test was performed by measuring both sides.

CONTACTS AND LOCATIONS:
Overall Officials: Beyza YAZGAN DAĞLI, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Central, Turkey (Türkiye)